CLINICAL TRIAL: NCT03020888
Title: A Prospective, Open Label, Post Marketing Study of Magseed and Sentimag in Patients Undergoing Surgical Excision of a Breast Lesion That Requires Preoperative Radiographic Localization
Brief Title: Magseed Magnetic Marker Localization
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Endomagnetics Inc (Industry)
Collaborators: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Organization: Endomagnetics Ltd. (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: US-002; NCT03019445 (obsolete NCT alias)
Record Dates: First submitted 2017-01-10; First posted 2017-01-13 (Estimated); Results first posted 2021-01-15 (Actual); Last update posted 2021-02-04 (Actual); Status verified 2021-01

CONDITIONS: Disorders of Breast; Breast Lesions
MeSH Terms: conditions — Breast Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Magseed and Sentimag (Experimental): Magseed marker deployed to mark a breast lesion under imaging guidance up to 30 days prior to surgery.
  Marker located during surgery using the Sentimag system, and removed with the lesion.
  Interventions: Device: Magseed and Sentimag

INTERVENTIONS:
Device: Magseed and Sentimag — Magseed marker and Sentimag probe for lesion localization

SUMMARY:
The purpose of this post-marketing study is to provide prospective evidence that the Magseed and Sentimag® is effective for lesion localization in patients undergoing surgical excision of a breast lesion and to summarize measures of product safety and performance.

DETAILED DESCRIPTION:
This is a post-market, prospective, open label, single arm study of Magseed and Sentimag in patients undergoing surgical excision of a breast lesion.

Subjects will have the Magseed marker deployed under imaging guidance up to thirty days prior to surgery.

The Magseed marker will be localized using the Sentimag system during surgery and removed with the lesion.

After the lumpectomy procedure, subjects will be evaluated for safety and patient reported outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with a breast lesion requiring image-guided localization prior to excision.
* Subjects aged 18 years or more at the time of consent.

Exclusion Criteria:

* The subject is pregnant or lactating.
* Subject has pacemaker or other implantable device in the chest wall.
* Subject has current active infection at the implantation site in the breast (per investigatordiscretion)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2018-02 (Actual); Study Completion 2018-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kelly Hunt, MD, Principal Investigator — MD Anderson
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Magseed and Sentimag: Magseed marker deployed to mark a breast lesion under imaging guidance up to 30 days prior to surgery.
  Marker located during surgery using the Sentimag system, and removed with the lesion.
  Magseed and Sentimag: Magseed marker and Sentimag probe for lesion localization
Period: Overall Study
Arm/Group | Magseed and Sentimag
Started | 120
Completed | 107
Not Completed | 13
Not completed — Physician Decision | 4
Not completed — Withdrawal by Subject | 6
Not completed — Insurance coverage | 2
Not completed — Lost to Follow-up | 1

BASELINE CHARACTERISTICS:
Arm/Group | Magseed and Sentimag
Number analyzed (Participants) | 107
Age, Continuous [Mean (Standard Deviation); unit: Years] | 60.73 (11.58)
Age, Continuous [Mean (Standard Deviation); unit: Years] | 60.73 (11.58)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 107
  Male | 0
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
BMI [Mean (Standard Deviation); unit: kg/m^2] | 28.83 (5.91)

OUTCOME MEASURES:

1. Primary Outcome: Percent of Participants With Retrieval of Index Lesion and Magseed
Description: Percent retrieval rate of the index lesion and Magseed in the initial excised specimen. This is defined as the number of subjects in whom the index lesion and Magseed are retrieved in the initial excised specimen divided by the total number of subjects undergoing surgery.
Time Frame: Time of surgery on average 16 minutes
Measure: Number; unit: percentage of participants
Arm/Group | Magseed and Sentimag
Number analyzed (Participants) | 107
percentage of participants | 100

2. Secondary Outcome: Number of Device Related Adverse Events
Description: Rates of device-related adverse events and device-related serious adverse events
Time Frame: 8 weeks
Measure: Number; unit: Number of device related adverse events
Arm/Group | Magseed and Sentimag
Number analyzed (Participants) | 107
Number of device related adverse events | 0

3. Secondary Outcome: Percent of Participants With Radiological Ease of Placement Rated as Very Easy, or Fairly Easy
Description: Radiologist were asked to rate ease of marker placement graded from Very easy, Fairly Easy & Difficult after each marker placement.
Time Frame: At the time of marker deployment on average 8.39 minutes
Measure: Number; unit: % Participants
Arm/Group | Magseed and Sentimag
Number analyzed (Participants) | 107
% Participants | 98

4. Secondary Outcome: Percentage of Markers With Radiological Placement Accuracy Measured as <5mm to Lesion
Description: Success rate of Magseed placement relative to the lesion (placement accuracy) measured as <5mm to lesion; 5-10mm to lesion; >10 mm to the target
Time Frame: At time of marker deployment on average 8.39 minutes
Population: 107 participants had 124 markers placed
Measure: Number; unit: percentage of markers
Units Other Than Participants: Markers
Arm/Group | Magseed and Sentimag
Number analyzed (Participants) | 107
Number analyzed (Markers) | 124
percentage of markers | 95.16

5. Secondary Outcome: Percentage of Participants With Re-excision
Description: Overall re-excision rate and re-excision rate necessary to remove the Magseed or targeted lesion
Time Frame: During surgery on average 16 minutes
Population: malignant breast lesions
Measure: Number; unit: percentage of participants
Arm/Group | Magseed and Sentimag
Number analyzed (Participants) | 98
percentage of participants | 9

6. Secondary Outcome: Percent of Participants With Surgical Ease of Localization - Rated Fairly or Very Easy
Description: Surgeon rated ease of localization during surgery assessed for each procedure as either very easy, fairly easy, fairly difficult, difficult, unable to localise
Time Frame: At time of surgery on average 16 minutes
Measure: Number; unit: percentage of participants
Arm/Group | Magseed and Sentimag
Number analyzed (Participants) | 107
percentage of participants | 86.9

7. Secondary Outcome: Surgical Localization - Duration of Localization
Description: Duration of the lumpectomy procedure, time taken to remove the lesion
Time Frame: At time of surgery on average 16 minutes
Measure: Mean (Full Range); unit: minutes
Arm/Group | Magseed and Sentimag
Number analyzed (Participants) | 107
minutes | 5 [1 to 45]

8. Secondary Outcome: Percentage of Participants With Marker Retrieval Rated as Fairly or Very Easy
Description: Pathologist rated ease of marker identification and retrieval as: 1) Unable to retrieve 2) Difficult 3) Fairly difficult 4)fairly easy 5) very easy
Time Frame: On the day of surgery
Measure: Number; unit: percentage of participants
Arm/Group | Magseed and Sentimag
Number analyzed (Participants) | 107
percentage of participants | 96

ADVERSE EVENTS:
Time Frame: Adverse vents data was captured from the time the Magseed was implanted to 8 weeks after it was surgically removed during the index procedure
Arm/Group | Magseed and Sentimag
All-Cause Mortality (participants affected / at risk) | 0/107
Serious Adverse Events (participants affected / at risk) | 0/107
Other Adverse Events (participants affected / at risk) | 0/107

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2016-12-30): https://cdn.clinicaltrials.gov/large-docs/88/NCT03020888/Prot_000.pdf
  • Statistical Analysis Plan (2018-06-24): https://cdn.clinicaltrials.gov/large-docs/88/NCT03020888/SAP_001.pdf